CLINICAL TRIAL: NCT02877160
Title: A Phase 1, Single-Center, Randomized, Open-Label, Single-Dose, Crossover Study to Assess the Pharmacokinetics, Including Food Effect, of AL-794 Formulations in Healthy Subjects
Brief Title: A Study to Assess the PK of AL-794 Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AL-794-803
Record Dates: First submitted 2016-07-11; First posted 2016-08-24 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — sfericase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Reference Formulation Fasted (Experimental): 150 mg of AL-794 study drug in suspension dosed in a fasted condition
  Interventions: Drug: AL-794 suspension
- Test Formulation Fasted (Experimental): 150 mg of AL-794 tablet formulation (3 x 50 mg tabs) dosed in a fasted condition
  Interventions: Drug: AL-794 tablet
- Test Formulation Fed (Experimental): 150 mg of AL-794 tablet formulation (3 x 50 mg tabs) dosed in a fed condition
  Interventions: Drug: AL-794 tablet

INTERVENTIONS:
Drug: AL-794 suspension
  Arms: Reference Formulation Fasted
Drug: AL-794 tablet
  Arms: Test Formulation Fasted; Test Formulation Fed

SUMMARY:
This study is a single-center, randomized, open-label crossover study to assess the pharmacokinetics and food effect of AL-794 formulations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written consent.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned.
3. Subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests and ECG.
4. Male or female, 18-60 years of age.
5. Body mass index (BMI) 18-30 kg/m2, inclusive. The minimum weight is 50 kg.
6. A female subject is eligible to participate in this study if she is of non-childbearing potential or postmenopausal.
7. If male, subject is surgically sterile or practicing acceptable forms of birth control until 90 days after the end of the study. Males must agree to refrain from sperm donation from check-in through 90 days after dosing.

Exclusion Criteria:

1. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 90 days after their last dose of study drugs.
2. Clinically significant laboratory abnormalities or abnormalities which are deemed to interfere with the ability to interpret study data.
3. Creatinine clearance of less than 60 mL/min (MDRD).
4. Total bilirubin, ALT, AST, or Alkaline Phosphatase >1.2×ULN (documented Gilbert's permitted).
5. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator and/or Sponsor's Medical Monitor.
6. Positive screening test for influenza, hepatitis A, B, C or HIV serology.
7. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
8. Participation in an investigational drug trial or having received an investigational vaccine within 3 months or 5 half-lives (whichever is longer) prior to study medication.
9. Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (eg, torsade de pointes), pre-existing sinus node disease, (incomplete) AV block, heart failure, or sudden cardiac death; or a corrected QT interval (QTcF or QTcB) >450 milliseconds for male subjects and >470 milliseconds for female subjects at the screening visit.
10. Clinically significant blood loss or elective blood donation of significant volume (ie, >500 mL) within 90 days of first dose of study drug; >1 unit of plasma within 7 days of first dose of study drug.
11. Clinically significant abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range, per local standards (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest) which are considered clinically significant. One repeat measurement after an additional 5 minutes of rest is permitted in one visit day.
12. Evidence of clinically significant infection within 2 weeks prior to admission.
13. Unwilling to abstain from alcohol for at least 1 week prior to the start of dosing through the Study Completion visit.
14. History of regular alcohol intake >14 units per week of alcohol for females and >21 units per week for males (one unit is defined as 8 g alcohol) within 3 months of the screening visit.
15. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening or Day 1.
16. History of tobacco use or used nicotine-containing products within 3 months of the screening visit.
17. The subject has a positive prestudy drug screen.
18. The use of concomitant medications, including prescription, over the counter medications, herbal medications, inducers or inhibitors of CYP enzymes, glucuronidation or drug transporters (including P-glycoprotein and OATP1B1) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. Occasional use of paracetamol, or its equivalent, is permitted.
19. Exposure to more than 4 new investigational entities within 12 months prior to the first dosing day.
20. Hypersensitivity to the active substances or to any of the excipients of AL-794, or prior dosing with AL-794.
21. Unwillingness or inability to comply with the study protocol for any other reason.
22. Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator or employees of Johnson & Johnson.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time of dosing to infinity (AUC0-inf) of ALS-033719 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions. | From Day 1 (Prior to dosing) to Day 14

SECONDARY OUTCOMES:
Safety as determined by AEs | From screening to Day 14
Safety as determined by Clinical lab results | From screening to Day 14
Safety as determined by 12-lead ECGs | From screening to Day 14
Safety as determined by Vital signs | From screening to Day 14
Safety as determined by Physical examinations | From screening to Day 14
Maximum observed concentration (Cmax) of ALS-033719 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions. | From Day 1 (Prior to dosing) to Day 14
Area under the concentration-time curve from time of dosing to last quantifiable concentration (AUC0-last) of ALS-033719 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions. | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: time of the maximum concentration (tmax) | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: terminal elimination half-life (t1/2) | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: Cmax | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: tmax | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: t1/2 | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: AUC0-inf | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033927 in plasma following single dose administration of test formulation and reference formulation of AL-794 under fasted conditions: AUC0-last | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033719 and ALS-033927 in plasma after a single oral dose of test formulation under fed conditions: Cmax | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033719 and ALS-033927 in plasma after a single oral dose of test formulation under fed conditions: Tmax | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033719 and ALS-033927 in plasma after a single oral dose of test formulation under fed conditions: AUC 0-inf | From Day 1 (Prior to dosing) to Day 14
PK parameters of ALS-033719 and ALS-033927 in plasma after a single oral dose of test formulation under fed conditions: AUC 0-last | From Day 1 (Prior to dosing) to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, Principal Investigator — HMR
Locations (1):
- Hammersmith Medicines Research Ltd (HMR), London, United Kingdom